CLINICAL TRIAL: NCT01463384
Title: MRI and MRS Diagnosis and Treatment Monitoring of Alzheimer's Disease With Novel Therapy
Brief Title: Minocycline in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huntington Medical Research Institutes (Other)
Responsible Party: Principal Investigator, Brian D. Ross, MD, Director, MR Unit, Huntington Medical Research Institutes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LKW-AB34
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Neuroinflammation; Mild Cognitive Impairment; Alzheimer's Disease; Minocycline
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Neuroinflammatory Diseases; cyclopia sequence | interventions — Minocycline; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Active Comparator): Subjects will be administered 50mg minocycline twice daily.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — 50mg, twice daily for 6 months.
  Other Names: Tetracycline

SUMMARY:
Cognitively normal individuals, patients with Mild Cognitive Impairment (MCI) or Alzheimer's Disease (AD) will undergo clinical screening, neuropsychological tests, blood and urine analyses, quantitative magnetic resonance imaging (MRI) and proton (1H ) and carbon 13 (13C) magnetic resonance spectroscopy (MRS). Each individual will receive minocycline oral administration for 4 weeks initially, after which MRI, MRS and neuropsychological results will be recorded. If no adverse side effects occur, subjects will continue minocycline administration for an additional 5 months.

DETAILED DESCRIPTION:
In the course of on-going trials of novel MRI procedures for Neurological Diagnosis, the investigators have established non-invasive BIOMARKERS (Note: Biomarkers are objective Laboratory tests used in, but not replacing Clinical diagnostic criteria of any disease,in this case age-related dementia of the Alzheimer type and its pre-clinical forms including Mild Cognitive Impairment - MCI) which significantly assist in the Diagnosis of Alzheimer's Disease. MRS, rather like blood tests which are applied for screening and exclusion of medical disorders, provides a pattern of brain chemicals from which this and many other diagnoses have become available (see: Magnetic Resonance Spectroscopy in Neurological Diagnosis: E.R Danielsen and B.D. Ross, Marcel Dekker New York, 1999). Diagnosis of Alzheimer's Disease has hitherto been exclusively a clinical diagnosis, made on the basis of non-specific tests by the treating physician/neurologist. Furthermore, treatments have been of limited efficacy so that the pressure for conclusive diagnosis or an objective characterization of disease progression (or better, regression) has not been a priority. This conservative approach to Alzheimer's Disease changed in 2010 with the Report of National Institutes of Aging. First: The failures of treatment have been ascribed to introduction only in patients with advanced disease ("dementia"). Second: A preliminary form of AD, known as pre-clinical or Mild Cognitive Impairment, has been recognized, distinct from, and generally earlier in the disease course. Third: A new set of diagnostic criteria, which include objective 'biomarkers', from cerebrospinal fluid, genetic and imaging analyzes, has been accepted by the Expert Panel. Finally, Clinical trials of existing and new drugs for Alzheimer's Disease are expected to yield better results if initiated earlier - in the pre-clinical phase - and the outcomes evaluated by the earlier changes in an approved panel of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal elderly subjects between the ages of 55-90 and patients aged 55 - 90 years who have mild cognitive impairment (MCI) or clinically defined Alzheimer's disease.

Exclusion Criteria:

* Any person with medical devices such as cardiac pacemakers/defibrillators or neuro-implants as they are contra-indications for MRI/MRS exam.
* Since the effects of MRI are unknown to the fetus or unborn child, any person who is or may be pregnant will be excluded from the study.
* History of known allergy or intolerance to minocycline or any other tetracycline
* Impaired renal function (plasma Creatinine) or blood urea nitrogen (BUN) levels exceeds twice normal upper limit which can result in higher serum levels of tetracycline, azotemia, hyperphosphatemia and acidosis.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Ross, Principal Investigator — Huntington Medical Research Institutes
Locations (1):
- Huntington Medical Research Institutes, Pasadena, California, United States

REFERENCES:
- See also: Related Info — http://www.hmri.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from local physicians, through Clinical Trials website and the AD association.
Groups:
- Minocycline: Subjects were administered 50mg minocycline twice daily for 6 months
Period: Overall Study
Arm/Group | Minocycline
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Minocycline: Subjects administered 50mg minocycline twice daily for 6 months
Arm/Group | Minocycline
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: RBANS is a brief neurocognitive battery with four alternate forms, measuring immediate and delayed memory, attention, language, and visuospatial skills. RBANS was developed as a stand-alone "core" battery for the detection and neurocognitive characterization of dementia and as a brief neurocognitive battery for the detection and tracking of neurocognitive deficits in a variety of disorders. (Reference: http://rbans.com/)
  Qualitative Description of Index Scores:
  Index Score Classification 130 and above Very Superior 120-129 Superior 110-119 High Average 90-109 Average 80-89 Low Average 70-79 Borderline 69 and below Extremely Low
  Psychometric range for RBANS:
  AD 0 - 77 MCI 78 - 99 Normal > 100
  Range of scores: Minimum = 0, Maximum = 130
  Values are reported below for Baseline, averaged for 1-3 months, and averaged for 4-6 months during minocycline administration.
Time Frame: Baseline values, 1-3 Months Values (averaged), 4-6 Months Values (averaged)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Minocycline AD: Alzheimer subjects who were administered 50mg minocycline twice daily.
- Minocycline MCI: Mild cognitively impaired subject who was administered 50mg minocycline twice daily.
- Minocycline NC: Normal control subjects who were administered 50mg minocycline twice daily.
Arm/Group | Minocycline AD | Minocycline MCI | Minocycline NC
Number analyzed (Participants) | 4 | 1 | 8
units on a scale
  Baseline Values | 49 (8) | 81 | 106 (13)
  Averaged Values for Months 1-3 | 32.5 (3.4) | 58.7 | 108.4 (26)
  Averaged Values for Months 4-6 | 32.9 (4.2) | 63.8 | 123.6 (37.1)

2. Primary Outcome: Hippocampal Volumes Measured in Three Groups: Alzheimer Disease (AD), Mild Cognitive Impairment (MCI) and Normal, Age-matched Controls (NC).
Description: Using magnetic resonance images acquired, hippocampal volume was measured monthly for 6 months.
  Normal range for hippocampal volume in aged-matched controls is 6.6 - 8.8 cm^3.
  Values are reported below for Baseline, averaged for 1-3 months, and averaged for 4-6 months during minocycline administration.
Time Frame: Baseline values, 1-3 Months Values (averaged), 4-6 Months Values (averaged)
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Minocycline AD | Minocycline MCI | Minocycline NC
Number analyzed (Participants) | 4 | 1 | 8
cm^3
  Baseline Values | 5.49 (1.14) | 6.35 | 6.98 (1.18)
  Averaged Values for Months 1-3 | 5.42 (1.06) | 6.30 | 6.92 (0.48)
  Averaged Values for Months 4-6 | 4.94 (1.2) | 7.60 | 6.82 (0.45)

3. Primary Outcome: Biomarker NAA/mI Measured in Three Groups: Alzheimer Disease (AD), Mild Cognitive Impairment (MCI) and Normal, Age-matched Controls (NC)
Description: It has been demonstrated in numerous studies over the past decade that magnetic resonance spectroscopy (MRS) can be used for the diagnosis of Alzheimer's disease. By measuring an area within the posterior cingulate gyrus, one can obtain a biochemical signature of that region in AD whereby NAA is reduced and mI is increased.
  These two biomarkers, N-acetylaspartate (NAA, a neuronal marker) and myo-inositol (mI, a glial marker) were quantified and then used to calculate NAA/mI (an index currently widely used for AD and MCI diagnosis).
  Scale of MRS biomarkers for aged-matched controls: NAA = 1.43, mI = 0.60, NAA/mI = 2.38. Any value lower than NAA/mI of 2.38 are considered not normal.
  Values are reported below for Baseline, averaged for 1-3 months, and averaged for 4-6 months during minocycline administration.
Time Frame: Baseline values, 1-3 Months Values (averaged), 4-6 Months Values (averaged)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Minocycline AD | Minocycline MCI | Minocycline NC
Number analyzed (Participants) | 4 | 1 | 8
Ratio
  Baseline Values | 1.69 (0.38) | 1.87 | 2.42 (0.08)
  Averaged Values for Months 1-3 | 1.78 (0.61) | 1.80 | 2.44 (0.26)
  Averaged Values for Months 4-6 | 1.84 (0.61) | 2.08 | 2.47 (0.41)

ADVERSE EVENTS:
Time Frame: 7 months
Description: No adverse events were reported.
Groups:
- Minocycline: No adverse events were reported in any subjects who were taking minocycline. All subjects underwent monthly blood tests to monitor alanine transaminase and blood urea nitrogen levels.
Arm/Group | Minocycline
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No